CLINICAL TRIAL: NCT05047497
Title: Ventilatory Functions, Oxygen Saturation, and Quality of Life Response to Long Time Cement Dust Exposure
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ramy Salama Draz, Principal Investigator, Cairo University
Other Study IDs: Cairo
Record Dates: First submitted 2020-09-04; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Occupational Diseases
MeSH Terms: conditions — Occupational Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- less than 10 years working: workers who work in cement factories in a period of time less than 10 years
  Interventions: Diagnostic Test: questionaire and ventilatory function test
- from 10-15 years working: workers who work in cement factories in a period of time from 10-15 years
  Interventions: Diagnostic Test: questionaire and ventilatory function test
- more than 15 years working: workers who work in cement factories in a period of time more than 15 years
  Interventions: Diagnostic Test: questionaire and ventilatory function test

INTERVENTIONS:
Diagnostic Test: questionaire and ventilatory function test — we assessed the arterial blood gases and the ventilatory functions and quality of life of whole three groups

SUMMARY:
Thousands of people are working daily in a dusty environment. Many studied reported respiratory symptoms and ventilatory disorders among Factory workers who exposed to cement dust. But the evidence for respiratory effect and daily activities over a long time of cement dust exposure has not been conclusive

DETAILED DESCRIPTION:
A total of 49 subjects working in a cement production factory were assessed and divided into three groups according to the total period of work exposure. Groupe A (18 subjects) with work period < 10 years, group B (13 subjects) with work period 10-15 years, group C (18 subjects) with work period > 15 years. The ventilatory functions, oxygen saturation, and quality of life were assessed in the three groups. RESULTS: The study results revealed a statistically significant difference between the three groups in the mean values of FVC (%), FEV1/FVC (%), SPO2.

ELIGIBILITY:
Inclusion Criteria:

* The ages were between 25 to 50 years old.
* the body mass index ranged from (18,5 - 29,9) kg/m2.

Exclusion Criteria:

* Age less than 25 or more 50.
* Any chronic diseases
* severe musculoskeletal and cardiopulmonary disorders and
* Class III Obesity (35-39.9 kg/m 2) or more

Ages: 25 Years to 50 Years | Sex: Male
Age Groups: Adult
Study Population: Out of sixty persons who were assigned to this study, a total of 49 subjects (group 1 n = 18, group 2 n = 13 and group 3 n = 18) completed the study (Fig. 1).
  In all groups, A, B and, C; height and weight scale were obtained for calculating BMI. The distribution of smokers between different age groups was measured (table ) The pulmonary function tests were performed to evaluate the capacity and volume of the lungs among the participants. Spirometry measurements, including FVC, FEV1, ratio of FEV1 to FVC (FEV1/FVC), forced expiratory flow 25-75% (FEF 25-75%), and peak expiratory flow (PEF
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
The ventilatory functions | 8 months
  ventilatory function tests were used to assess FVC (%), FEV1/FVC (%),PEF (%), FEV1 (%)
oxygen saturation | 8 months
  measuring oxygen saturation using SPo2
quality of life were assessed | 8 months
  the mean values of the physical functioning item and energy/fatigue item in the quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Cairo, Egypt